CLINICAL TRIAL: NCT01747850
Title: Sativex Associated With Behavioral-relapse Prevention Strategy as Treatment for Cannabis Dependence
Brief Title: Sativex and Behavioral-relapse Prevention Strategy in Cannabis Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Bernard Le Foll, Head, Translational Addiction Research Laboratory, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 144/2011; R21DA031906 (NIH)
Record Dates: First submitted 2012-12-07; First posted 2012-12-12 (Estimated); Results first posted 2017-10-02 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-07

CONDITIONS: Cannabis Dependence
MeSH Terms: conditions — Marijuana Abuse | interventions — Cognitive Behavioral Therapy; nabiximols; Dronabinol; Cannabidiol; Ethanol; Color

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sativex (Experimental): Intervention consist on Sativex Spray (Δ9-tetrahydrocannabinol/cannabidiol). Study subjects will be randomized in blocks of ten to one of the two groups (Sativex vs. placebo) in a double blind manner. There will be a gradual increase of the maximal allowed dose starting at five sprays per day for the first two days and increasing of five sprays per day until reaching the max number of 42 sprays per day at the end of week 2. There will be a total of 12 weeks of drug exposure. All participants will receive a combination of pharmacotherapy (Sativex or Placebo) associated with a weekly intervention of combined Motivational Enhancement/Cognitive Behavioral Therapy.
  Interventions: Behavioral: Motivational Enhancement/Cognitive Behavioral Therapy; Drug: Sativex
- Placebo spray (Placebo Comparator): Participants will receive a combination of Placebo spray associated with a weekly intervention of combined Motivational Enhancement Therapy and Cognitive Behavioral Therapy
  Interventions: Behavioral: Motivational Enhancement/Cognitive Behavioral Therapy; Drug: Placebo spray
- Pilot Study (Experimental): The first five subjects will be treatment-seekers that fit our inclusion/exclusion criteria and that will be treated open-label. These subjects will be instructed to use the Sativex Spray according to the induction schedule provided above. These first subjects will allow us to determine if our schedule for dosing is appropriate for the subsequent phase of the study.
  Interventions: Behavioral: Motivational Enhancement/Cognitive Behavioral Therapy; Drug: Sativex

INTERVENTIONS:
Behavioral: Motivational Enhancement/Cognitive Behavioral Therapy — All participants will receive a combination of pharmacotherapy (Sativex or Placebo) associated with a weekly intervention of combined Motivational Enhancement Therapy and Cognitive Behavioral Therapy.
Drug: Sativex — Study subjects will gradually increase the maximal allowed dose of Sativex starting at five sprays per day for the first two days and increasing of five sprays per day until reaching the max number of 42 sprays maximal per day at end of week 2 (Day 11). The target quit date will be set at Day 21 (but subjects will be allowed to stop using cannabis before if they are willing and able to). The medication treatment phase will then be continued for an additional 9 weeks (the last week will be a reduction phase with the use of Spray that will be decreased by 50% to avoid abrupt withdrawal). Then exposure to medications will be stopped (so there will be a total of 12 weeks medication treatment exposure).
  Other Names: delta-9-tetrahydrocannabinol and cannabidiol
  Arms: Pilot Study; Sativex
Drug: Placebo spray — Study subjects will gradually increase the maximal allowed dose of Placebo starting at five sprays per day for the first two days and increasing of five sprays per day until reaching the max number of 42 sprays maximal per day at end of week 2 (Day 11). The target quit date will be set at Day 21 (but subjects will be allowed to stop using cannabis before if they are willing and able to). The Placebo treatment phase will then be continued for an additional 9 weeks (the last week will be a reduction phase with the use of Placebo Spray that will be decreased by 50%). Then exposure to Placebo will be stopped (so there will be a total of 12 weeks Placebo treatment exposure).
  Other Names: Ethanol,propylene glycol,and peppermint oil with colors
  Arms: Placebo spray

SUMMARY:
The purpose of this study is assess Sativex as a treatment for Cannabis dependence. Initially a pilot study will be conducted in five subjects seeking treatment for cannabis dependence to ensure that our planned self-titration regimen is appropriate using Sativex. This phase will be open label, with no placebo control. Then, there will be a twelve-week, double-blind, placebo-controlled study in male and female subjects seeking treatment for cannabis dependence (n=40). All participants will receive a combination of pharmacotherapy (Sativex Spray or Placebo Spray) associated with a weekly intervention of combined Motivational Enhancement Therapy and Cognitive Behavioral Therapy (MET/CBT). The subjects will have to come daily to the centre to assess usage of medication. Following the medication phase, participants will have a follow-up weekly for another four weeks and then monthly until the 6 month follow up visit after the target quit date. The investigators are planning to enroll 45 subjects over the two-year period.

DETAILED DESCRIPTION:
In the pilot study subjects will be treated with SATIVEX® (THC/cannabidiol combination in a buccal spray) using the same approach as outlined below for the randomized controlled trial. In the twelve-week, double-blind, placebo-controlled study visits will occur weekly during the medication phase of the study. The medication will be self-titrated over three weeks and a target quit date will be set up at Day 21. There will be a total of 12 weeks of drug exposure. Throughout these 12-weeks, all participants will receive a combination of pharmacotherapy (Sativex Spray or Placebo Spray) associated with a weekly intervention of combined Motivational Enhancement Therapy and Cognitive Behavioral Therapy (MET/CBT) in accordance with the intervention practices shown to be effective in treatment of cannabis dependence. The intervention will be adapted from the Brief Counselling for Marijuana Dependence manual published by the Substance Abuse and Mental Health Services Administration (SAMHSA). At each study visit, vital signs and self-report ratings will be collected. In addition, the subjects will have to come daily to the centre to assess medication usage and will be asked to provide urine sample (two times weekly) and blood sample weekly. As there may be compliance issues, a contingency management approach will be also implemented.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female (gender to be analyzed as a covariate)
* Understand and willing to comply with study requirements and restrictions
* Willing to use appropriate contraceptive method throughout the study
* Otherwise healthy as judged by investigator based on medical history, physical exam, vitals, ECG and labs
* DSM-IV criteria for current marijuana dependence
* Report marijuana as primary drug of abuse
* Report using marijuana at least 5 days a week for at least one month
* Have marijuana positive urine drug screen
* Treatment seeking cannabis smoker
* Smoke less than or equal to the equivalent of 4 joints per day (or four grams per day if participants smokes cannabis in other forms)

Exclusion Criteria:

* Meets DSM-IV criteria for a current axis I disorder including substance use disorder other than cannabis, nicotine or caffeine dependence.
* First-degree relative with schizophrenia
* History of seizures
* History of cardiovascular disease
* History of pulmonary disease such as asthma, COPD
* Clinically significant pathology in oral cavity and poor oral hygiene
* Known sensitivity to dronabinol, cannabidiol, propylene glycole, ethanol or peppermint oil (used in SATIVEX® buccal spray)
* Unstable medical conditions
* Pregnant or breast-feeding
* Currently taking psychotropic medication with benefit for any other illness than treatment of insomnia,
* Holding a job that involves driving, operating heavy machines

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Le Foll, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang R, Trigo JM, Le Foll B. Effects of sub-chronic nabiximols on biological markers of individuals undergoing a clinical trial for the treatment of cannabis use disorder. Am J Transl Res. 2023 Aug 15;15(8):5228-5238. eCollection 2023. PMID 37692969
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital, fully affiliated with the University of Toronto, and a PAHO/WHO Collaborating Centre — http://www.camh.net/research

RESULTS

PARTICIPANT FLOW:
Groups:
- Pilot Study: The first five subjects will be treatment-seekers that will be treated open-label. These first subjects will allow us to determine if our schedule for dosing is appropriate for the subsequent phase of the study.
  Motivational Enhancement/Cognitive Behavioral Therapy: All participants will receive a combination of pharmacotherapy (Sativex) associated with a weekly intervention of combined Motivational Enhancement Therapy and Cognitive Behavioral Therapy.
  Sativex: Study subjects will gradually increase the maximal allowed dose of Sativex starting at five sprays per day for the first two days and increasing of five sprays per day until reaching the max number of 42 sprays maximal per day at end of week 2 (Day 11). The medication treatment phase will then be continued for an additional 9 weeks (the last week will be a reduction phase with the use of Spray that will be decreased by 50% to avoid abrupt withdrawal).
- Sativex: Intervention consist on Sativex Spray (Δ9-tetrahydrocannabinol/cannabidiol). Study subjects will be randomized in blocks of ten to one of the two groups (Sativex vs. placebo) in a double blind manner. There will be a gradual increase of the maximal allowed dose starting at five sprays per day for the first two days and increasing of five sprays per day until reaching the max number of 42 sprays per day at the end of week 2. There will be a total of 12 weeks of drug exposure (the last week will be a reduction phase with the use of Spray that will be decreased by 50% to avoid abrupt withdrawal). All participants will receive a combination of pharmacotherapy (Sativex or Placebo) associated with a weekly intervention of combined Motivational Enhancement/Cognitive Behavioral Therapy.
- Placebo Spray: Participants will receive a combination of Placebo spray associated with a weekly intervention of combined Motivational Enhancement Therapy and Cognitive Behavioral Therapy
  Placebo spray: Study subjects will gradually increase the maximal allowed dose of Placebo starting at five sprays per day for the first two days and increasing of five sprays per day until reaching the max number of 42 sprays maximal per day at end of week 2 (Day 11). The Placebo treatment phase will then be continued for an additional 9 weeks (the last week will be a reduction phase with the use of Placebo Spray that will be decreased by 50%). Then exposure to Placebo will be stopped (so there will be a total of 12 weeks Placebo treatment exposure).
Period: Overall Study
Arm/Group | Pilot Study | Sativex | Placebo Spray
Started | 5 | 20 | 20
Completed | 4 | 13 | 14
Not Completed | 1 | 7 | 6

BASELINE CHARACTERISTICS:
Groups:
- Sativex: Intervention consist on Sativex Spray (Δ9-tetrahydrocannabinol/cannabidiol). There will be a gradual increase of the maximal allowed dose starting at five sprays per day for the first two days and increasing of five sprays per day until reaching the max number of 42 sprays per day at the end of week 2. There will be a total of 12 weeks of drug exposure associated with a weekly intervention of combined Motivational Enhancement/Cognitive Behavioral Therapy.
  Sativex: Study subjects will gradually increase the maximal allowed dose of Sativex starting at five sprays per day for the first two days and increasing of five sprays per day until reaching the max number of 42 sprays maximal per day at end of week 2 (Day 11). The medication treatment phase will then be continued for an additional 9 weeks (the last week will be a reduction phase with the use of Spray that will be decreased by 50% to avoid abrupt withdrawal).
- Placebo Spray: Participants will receive a combination of Placebo spray associated with a weekly intervention of combined Motivational Enhancement Therapy and Cognitive Behavioral Therapy
  Placebo spray: Study subjects will gradually increase the maximal allowed dose of Placebo starting at five sprays per day for the first two days and increasing of five sprays per day until reaching the max number of 42 sprays maximal per day at end of week 2 (Day 11). The Placebo treatment phase will then be continued for an additional 9 weeks (the last week will be a reduction phase with the use of Placebo Spray that will be decreased by 50%).
- Pilot Study: The first five subjects will be treatment-seekers that fit our inclusion/exclusion criteria and that will be treated open-label. These first subjects will allow us to determine if our schedule for dosing is appropriate for the subsequent phase of the study.
  All participants will receive a combination of pharmacotherapy (Sativex) associated with a weekly intervention of combined Motivational Enhancement Therapy and Cognitive Behavioral Therapy.
  Sativex: Study subjects will gradually increase the maximal allowed dose of Sativex starting at five sprays per day for the first two days and increasing of five sprays per day until reaching the max number of 42 sprays maximal per day at end of week 2 (Day 11). The medication treatment phase will then be continued for an additional 9 weeks (the last week will be a reduction phase with the use of Spray that will be decreased by 50% to avoid abrupt withdrawal).
- Total: Total of all reporting groups
Arm/Group | Sativex | Placebo Spray | Pilot Study | Total
Number analyzed (Participants) | 20 | 20 | 5 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 5 | 45
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 2 | 13
  Male | 15 | 14 | 3 | 32
Region of Enrollment [Number; unit: participants]
  Canada | 20 | 20 | 5 | 45

OUTCOME MEASURES:

1. Primary Outcome: Tolerability
Description: Assessment of tolerability will be determined by the number of subjects that withdrawal from the study due to SAEs.
Time Frame: six months
Measure: Count of Participants; unit: Participants
Groups:
- Sativex # of Participants That Withdrew Due SAE: Intervention consist on Sativex Spray (Δ9-tetrahydrocannabinol/cannabidiol). There will be a total of 12 weeks of drug exposure. All participants will receive a combination of pharmacotherapy (Sativex associated with a weekly intervention of combined Motivational Enhancement/Cognitive Behavioral Therapy.
- Placebo # of Participants That Withdrew Due SAE: Participants will receive a combination of Placebo spray associated with a weekly intervention of combined Motivational Enhancement Therapy and Cognitive Behavioral Therapy
- Pilot Study # of Participants That Withdrew Due SAE: The first five subjects will be treatment-seekers that fit our inclusion/exclusion criteria and that will be treated open-label. These subjects will be instructed to use the Sativex Spray according to the induction schedule provided above. These first subjects will allow us to determine if our schedule for dosing is appropriate for the subsequent phase of the study.
  Motivational Enhancement/Cognitive Behavioral Therapy: All participants will receive a combination of pharmacotherapy (Sativex or Placebo) associated with a weekly intervention of combined Motivational Enhancement Therapy and Cognitive Behavioral Therapy.
  Sativex: Study subjects will gradually increase the maximal allowed dose of Sativex starting at five sprays per day for the first two days and increasing of five sprays per day until reaching the max number of 42 sprays maximal per day at end of week 2 (Day 11). The target quit date will be set at Day 21 (but subjects will be allowed to stop using cannabis before if
Arm/Group | Sativex # of Participants That Withdrew Due SAE | Placebo # of Participants That Withdrew Due SAE | Pilot Study # of Participants That Withdrew Due SAE
Number analyzed (Participants) | 20 | 20 | 5
Participants | 0 | 0 | 0

2. Secondary Outcome: Cannabis Use (in Days)
Description: The percentage of days that participants self-reported use of cannabis over the study duration until 6 month follow-up will be assessed (i.e. smoking diary self-report)
Time Frame: six months
Measure: Mean (Standard Deviation); unit: percentage of days
Groups:
- Sativex % Days Use of Cannabis: Intervention consist on Sativex Spray (Δ9-tetrahydrocannabinol/cannabidiol). There will be a total of 12 weeks of drug exposure. All participants will receive a combination of pharmacotherapy (Sativex associated with a weekly intervention of combined Motivational Enhancement/Cognitive Behavioral Therapy.
- Placebo % Days Use of Cannabis: Participants will receive a combination of Placebo spray associated with a weekly intervention of combined Motivational Enhancement Therapy and Cognitive Behavioral Therapy
- Pilot % Days Use of Cannabis: The first five subjects will be treatment-seekers that fit our inclusion/exclusion criteria and that will be treated open-label.
Arm/Group | Sativex % Days Use of Cannabis | Placebo % Days Use of Cannabis | Pilot % Days Use of Cannabis
Number analyzed (Participants) | 20 | 20 | 5
percentage of days | 42.9 (7.7) | 47.1 (12.9) | 48.3 (22.5)

3. Secondary Outcome: Withdrawal
Description: Effect of Sativex on withdrawal symptom scores will be assessed using the Marijuana Withdrawal Checklist (MWC). Average Total score for the trial (6 months) is reported.
  Range 0 - 46. Higher scores indicate more severe symptoms associated with marijuana withdrawal.
Time Frame: six months
Measure: Mean (Standard Deviation); unit: Total Withdrawal score
Groups:
- Sativex Withdrawal: Intervention consist on Sativex Spray (Δ9-tetrahydrocannabinol/cannabidiol). There will be a total of 12 weeks of drug exposure. All participants will receive a combination of pharmacotherapy (Sativex associated with a weekly intervention of combined Motivational Enhancement/Cognitive Behavioral Therapy.
- Placebo Withdrawal: Participants will receive a combination of Placebo spray associated with a weekly intervention of combined Motivational Enhancement Therapy and Cognitive Behavioral Therapy
- Pilot Withdrawal: The first five subjects will be treatment-seekers that fit our inclusion/exclusion criteria and that will be treated open-label.
Arm/Group | Sativex Withdrawal | Placebo Withdrawal | Pilot Withdrawal
Number analyzed (Participants) | 20 | 20 | 5
Total Withdrawal score | 5.0 (4.7) | 5.1 (3.9) | 2.7 (2.5)

4. Secondary Outcome: Cannabis Craving
Description: Effect of Sativex on cannabis craving will be assessed using the Marijuana Craving Questionnaire (MCQ). Average Total score for the trial (6 months) is reported.
  Participants rate the 12 items using a 7-item Likert scale ranging from strongly disagree to strongly agree, and the total score ranges from 4 to 28 (subscales compulsivity (mean items 2, 7 and 10), emotionality (mean items 4, 6 and 9), expectancy (mean items 5, 11 and 12) and purposefulness (mean items 1, 3 and 8); total score is the sum for the 4 subscales). Higher scores indicate more severe craving for marijuana.
Time Frame: six months
Measure: Mean (Standard Deviation); unit: Total Craving Scores
Groups:
- Sativex Craving: Intervention consist on Sativex Spray (Δ9-tetrahydrocannabinol/cannabidiol). There will be a total of 12 weeks of drug exposure. All participants will receive a combination of pharmacotherapy (Sativex associated with a weekly intervention of combined Motivational Enhancement/Cognitive Behavioral Therapy.
- Placebo Craving: Participants will receive a combination of Placebo spray associated with a weekly intervention of combined Motivational Enhancement Therapy and Cognitive Behavioral Therapy
- Pilot Craving: The first five subjects will be treatment-seekers that fit our inclusion/exclusion criteria and that will be treated open-label.
Arm/Group | Sativex Craving | Placebo Craving | Pilot Craving
Number analyzed (Participants) | 20 | 20 | 5
Total Craving Scores | 8.2 (4.3) | 9.6 (5.7) | 9.5 (5.2)

5. Secondary Outcome: Cannabis Use (Grams)
Description: Amount of cannabis used in grams over the study duration until 6 month follow-up will be assessed
Time Frame: six months
Measure: Mean (Standard Error); unit: grams of cannabis
Groups:
- Sativex Cannabis Use (g): Intervention consist on Sativex Spray (Δ9-tetrahydrocannabinol/cannabidiol). There will be a total of 12 weeks of drug exposure. All participants will receive a combination of pharmacotherapy (Sativex associated with a weekly intervention of combined Motivational Enhancement/Cognitive Behavioral Therapy.
- Placebo Cannabis Use (g): Participants will receive a combination of Placebo spray associated with a weekly intervention of combined Motivational Enhancement Therapy and Cognitive Behavioral Therapy
- Pilot Cannabis Use (g): The first five subjects will be treatment-seekers that fit our inclusion/exclusion criteria and that will be treated open-label.
Arm/Group | Sativex Cannabis Use (g) | Placebo Cannabis Use (g) | Pilot Cannabis Use (g)
Number analyzed (Participants) | 20 | 20 | 5
grams of cannabis | 2.3 (0.76) | 3.5 (1.26) | 1.6 (1.48)

ADVERSE EVENTS:
Time Frame: 1 year, 10 months
Description: ADVERSE EVENT COLLECTION BY QUESTIONNAIRE DURING STUDY VISITS (SAFTEE)
Groups:
- Sativex: Intervention consist on Sativex Spray (Δ9-tetrahydrocannabinol/cannabidiol). There will be a gradual increase of the maximal allowed dose starting at five sprays per day for the first two days and increasing of five sprays per day until reaching the max number of 42 sprays per day at the end of week 2. There will be a total of 12 weeks of drug exposure.
  All participants will receive a combination of pharmacotherapy (Sativex ) associated with a weekly intervention of combined Motivational Enhancement Therapy and Cognitive Behavioral Therapy.
- Placebo Spray: Placebo spray: Study subjects will gradually increase the maximal allowed dose of Placebo starting at five sprays per day for the first two days and increasing of five sprays per day until reaching the max number of 42 sprays maximal per day at end of week 2 (Day 11). There will be a total of 12 weeks Placebo treatment exposure.
  Participants will receive a combination of Placebo spray associated with a weekly intervention of combined Motivational Enhancement Therapy and Cognitive Behavioral Therapy
- Pilot Study: The first five subjects will be treatment-seekers that will be treated open-label.
  Study subjects will gradually increase the maximal allowed dose of Sativex starting at five sprays per day for the first two days and increasing of five sprays per day until reaching the max number of 42 sprays maximal per day at end of week 2 (Day 11). There will be a total of 12 weeks medication treatment exposure).
  Motivational Enhancement/Cognitive Behavioral Therapy: All participants will receive a combination of pharmacotherapy (Sativex) associated with a weekly intervention of combined Motivational Enhancement Therapy and Cognitive Behavioral Therapy.
Arm/Group | Sativex | Placebo Spray | Pilot Study
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/5
Other Adverse Events (participants affected / at risk) | 16/20 | 18/20 | 4/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sativex (N=20) | Placebo Spray (N=20) | Pilot Study (N=5)
Insomnia (Nervous system disorders) | 11 | 8 | 3
Headache (Vascular disorders) | 4 | 10 | 3
Oro Mucal (Gastrointestinal disorders) | 2 | 2 | 2
Cold/Influenza (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 3
Cardiovascular (Cardiac disorders) | 0 | 2 | 0
Nightmare (General disorders) | 0 | 2 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 4 | 1
Pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Mood Disturbance (Psychiatric disorders) | 2 | 0 | 1
Decrease in Libido (Psychiatric disorders) | 0 | 3 | 0
Decreased appetite (General disorders) | 2 | 2 | 1
Nausea (Gastrointestinal disorders) | 2 | 6 | 2
Urinary Problems (Renal and urinary disorders) | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 1
Skin rashes (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Indigestion (Gastrointestinal disorders) | 0 | 0 | 1
Light Headedness (Cardiac disorders) | 0 | 0 | 1
excessive sweating (Nervous system disorders) | 0 | 2 | 1
Ringing in ears (General disorders) | 2 | 0 | 1
Walking up in the middle of night (Psychiatric disorders) | 0 | 0 | 1
Tiredness (General disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes